CLINICAL TRIAL: NCT02099214
Title: Estimation of Myocardial Iron Overload by 3 Tesla MRI and Cardiac Functional Consequences in Patients With HFE Hereditary Haemochromatosis. Pilot Study
Brief Title: Estimation of Myocardial Iron Overload by 3 Tesla MRI in HFE Hereditary Haemochromatosis
Acronym: HEMOCOEUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A01843-42
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Iron Overload; HFE-Associated Hereditary Hemochromatosis
Keywords: myocardial iron overload; HFE-Associated Hereditary Hemochromatosis; 3 Tesla MRI; cardiological strategy in haemochromatosis; congestive heart failure
MeSH Terms: conditions — Heart Failure | interventions — Electrocardiography; Iron; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with HFE hereditary haemochromatosis (Experimental): The patients (40) will undergo a medical examination in order to analyse their medical history, cardiovascular parameters and check inclusion and non-inclusion criterions.
  Then will be performed :
  * An electrocardiogram
  * Blood tests : iron and cardiac markers (serum iron, serum transferrin, transferrin saturation, serum ferritin, NT-proBNP), beta-hCG if needed, serum bank
  * A 3Tesla cardiac MRI repeated twice (in order to respect the reproducibility criterion)
  * A 3Tesla abdominal MRI
  * An echocardiography at rest.
  Interventions: Device: 3Tesla cardiac MRI; Device: Electrocardiogram (EKG); Biological: Iron and cardiac markers; Biological: Pregnancy test; Device: Echocardiography at rest; Device: 3Tesla abdominal MRI
- Healthy volunteers (Experimental): The healthy volunteers (10 men and 10 women) will undergo :
  * A urinary pregnancy test (if applicable)
  * A 3Tesla cardiac MRI repeated twice (in order to respect the reproducibility criterion)
  * An echocardiography at rest.
  Interventions: Device: 3Tesla cardiac MRI; Device: Echocardiography at rest; Biological: Urinary pregnancy test

INTERVENTIONS:
Device: 3Tesla cardiac MRI
Device: Electrocardiogram (EKG)
  Arms: Patients with HFE hereditary haemochromatosis
Biological: Iron and cardiac markers — Serum iron, serum transferrin, transferrin saturation, serum ferritin, NT-proBNP
  Arms: Patients with HFE hereditary haemochromatosis
Biological: Pregnancy test — Beta-hCG
  Arms: Patients with HFE hereditary haemochromatosis
Device: Echocardiography at rest — Transthoracic echocardiograph
Biological: Urinary pregnancy test
  Arms: Healthy volunteers
Device: 3Tesla abdominal MRI
  Arms: Patients with HFE hereditary haemochromatosis

SUMMARY:
Hereditary haemochromatosis (HHC) is a frequent disease in Brittany (5 to 7‰), responsible first for biological disorder in blood iron parameters and minor clinical disorders, before evolving to potential life-threatening consequences such as diabetes, liver cirrhosis and congestive heart failure.

The improvement of screening and treatments made those severe affections rare enough not to evaluate myocardial iron overload a systematic part of the starting check-up. Nonetheless this myocardial iron overload might have severe implications on cardiac function on a long term basis.

A single trial was conducted on limited number of patients with 1.5 Tesla MRI, which showed a myocardial iron overload (defined by a myocardium T2* value <20ms) in 19% of the subjects.

The main objective of this study is to precisely estimate cardiac iron overload in treatment naive patients with newly diagnosed HFE hereditary haemochromatosis with a 3 Tesla MRI, more sensitive than the 1.5 Tesla one, in order to later appreciate its correlation with cardiac morbidity in HHC.

DETAILED DESCRIPTION:
Since the wide use of phlebotomy was implemented the incidence of congestive heart failure in HHC became quite low. As such, the interest towards the initial diagnosis and cardiological follow-up has been lesser. A subclinical myocardial iron overload can nevertheless exist and eventually lead to functional consequences in the medium and long term if neglected, even evolve into heart failure and preserved ejection fraction.

The expected aftermath of this study is :

* The estimation of the frequency of myocardial iron overload measured by 3 Tesla MRI in patient with HFE hereditary haemochromatosis;
* The assessment of its consequences on heart function;
* The appreciation of a cardiological assessment strategy in patients with HFE hereditary haemochromatosis.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Adults older than 18 ;
* Newly diagnosed with HFE hereditary haemochromatosis by genetic testing (homozygous for the C283Y mutation on HFE gene);
* Treatment-naive;
* Showing a ferritin level higher than 200µg/l for women and higher than 300µg/L for men;
* Affiliated to French Social Security;
* Having given a written informed consent.

Healthy volunteers:

* Adults older than 18;
* Presenting all the following criterions:

  * Normal cardiovascular physical examination: no signs of cardiac insufficiency, no pathological cardiac murmur, normal EKG (regular sinus rhythm, no high degree AV nor ventricular blocks, no rhythm anomaly),
  * Body Mass Index <27 kg/m²,
  * Normal routine blood biology (blood count, MCV, serum iron, ferritin, transferrin saturation);
* Affiliated to French Social Security;
* Having given a written informed consent.

Exclusion Criteria:

Patients :

MRI-related criterions :

* Cardiac pacemaker or implanted defibrillator ;
* Non MRI-compatible prosthetic cardiac valve;
* Non MRI-compatible clips/stents/coils/etc.;
* Cochlear implant;
* Peripheral or neuronal stimulator;
* Intra-ocular or brain metallic foreign bodies , foreign body in the eyes' vicinity, shrapnel or firearm wound;
* Less than 4 weeks-old stents, less than 6 weeks-old osteosynthesis materials;
* Claustrophobia;
* Pumps, tattoos, permanent makeup, intrauterine device, patches;
* Non-removable metallic or magnetic material in the vicinity of the analysed field.

Other criterions :

* Haemodynamic instability / Acute respiratory insufficiency / Altered general status / Need for continuous monitoring incompatible wih MRI confines;
* Pregnancy, breast feeding;
* History of blood transfusion or iron supplementation;
* Blood donation in the last 3 months;
* Infection in the 7 days prior to the first visit;
* Stay in altitude (>1500m) in the past 2 months;
* Adults under legal protective regimen or deprived of liberty.

Healthy volunteers

* Alcohol abuse (>20g per day for women, >30g per day for men);
* Active tobacco intoxication or smoking cessation in the 6 last months;
* Personal cardiovascular medical history;
* Cardiovascular functional signs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Myocardial T2* values in haemochromatosis compared to healthy volunteers | Day 1
  Assessment of the percentage rate of patients presenting a lower T2* value than the baseline defined by the mean of T2* values measured in healthy volunteers with a 1 standard deviation margin.

SECONDARY OUTCOMES:
Mean T2 values in healthy volunteers and patients with HFE-related haemochromatosis | Day 1
  Comparison of the mean T2 values in healthy volunteers and patients with HFE-related haemochromatosis
Echocardiographic parameters of systolic and diastolic functions and myocardial deformation | Day 1
Myocardial T2 and T2* values in both groups | Day 1
Liver T2/T2* values | Day 1
  Correlation between liver T2/T2* and myocardial T2/T2*
Pancreas T2/T2* values | Day 1
  Correlation between pancreas T2/T2* and myocardial T2/T2*
Spleen T2/T2* values | Day 1
  Correlation between spleen T2/T2* and myocardial T2/T2*

CONTACTS AND LOCATIONS:
Overall Officials: Erwan DONAL, MD, PhD, Principal Investigator — Rennes University Hospital - Service de cardiologie et maladies vasculaires; Bruno LAVIOLLE, MD, PhD, Study Chair — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France